CLINICAL TRIAL: NCT06564012
Title: Wearable Cardiac Monitor to Enhance Detection of Arrhythmia Recurrence After Catheter Ablation of Atrial Fibrillation
Acronym: WEAR-AF
Status: Not yet recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 4513
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases; Stroke Prevention
Keywords: digital health; wearable technology; electrocardiography; remote monitoring; patient adherence
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The WEAR-AF study is a prospective, multicenter clinical trial designed to evaluate the efficacy of wearable technology in the detection, monitoring, and management of atrial fibrillation (AF). This study aims to assess how wearable devices, such as smartwatches equipped with electrocardiogram (ECG) capabilities, can be used to identify AF episodes, guide treatment decisions, and ultimately improve patient outcomes.

Participants will be individuals diagnosed with or at high risk for atrial fibrillation. The study will track the accuracy of AF detection, patient adherence to monitoring, and the impact on clinical outcomes, including stroke prevention, symptom management, and quality of life.

The findings from WEAR-AF are expected to contribute to the growing body of evidence supporting the integration of wearable technology into routine clinical practice for AF management, offering insights into its potential to enhance patient care and reduce healthcare costs.

DETAILED DESCRIPTION:
Study Description:

The WEAR-AF study is a prospective, multicenter clinical trial designed to evaluate the effectiveness and clinical utility of wearable technology in the detection, monitoring, and management of atrial fibrillation (AF). This study seeks to understand how wearable devices, particularly those with electrocardiogram (ECG) capabilities, can be integrated into routine clinical practice to enhance the early detection and continuous monitoring of AF, a common and potentially serious cardiac arrhythmia.

Background and Rationale:

Atrial fibrillation is a significant public health issue, associated with increased risks of stroke, heart failure, and other cardiovascular complications. Current guidelines emphasize the importance of early detection and continuous monitoring of AF to manage symptoms and prevent complications effectively. Wearable technology, such as smartwatches and fitness trackers equipped with ECG functions, has emerged as a promising tool for real-time AF detection and monitoring. However, the clinical efficacy, accuracy, and patient adherence associated with these devices require further investigation.

Objectives:

The primary objective of the WEAR-AF study is to evaluate the diagnostic accuracy of wearable ECG devices in detecting AF episodes compared to standard clinical practices, such as Holter monitoring and traditional ECGs. Secondary objectives include assessing the impact of continuous AF monitoring on clinical outcomes, including stroke prevention, symptom management, and patient quality of life. The study will also examine patient adherence to the use of wearable technology and its influence on healthcare utilization and costs.

Study Design:

WEAR-AF is a prospective, observational study that will enroll participants across multiple centers. Eligible participants include individuals diagnosed with AF or those at high risk for developing AF. Participants will be provided with wearable devices equipped with ECG capabilities and will be monitored over a specified period. The study will compare the AF detection rates of these wearable devices against standard diagnostic tools, evaluate the consistency of AF management with the wearable devices' data, and document any changes in clinical outcomes over time.

Endpoints:

Primary Endpoint:

Diagnostic accuracy of wearable ECG devices in detecting AF compared to standard methods.

Secondary Endpoints:

Impact of wearable ECG monitoring on stroke incidence and other cardiovascular events.

Changes in AF-related symptoms and quality of life as measured by validated questionnaires.

Patient adherence to the use of wearable technology for continuous AF monitoring.

Healthcare utilization and cost-effectiveness analysis.

Significance:

The WEAR-AF study aims to generate robust evidence on the role of wearable technology in managing AF. By providing insights into the accuracy, utility, and patient adherence to these devices, the study will contribute to the development of guidelines for the integration of wearable technology into clinical practice. The ultimate goal is to improve patient outcomes by enabling more timely and precise management of AF.

Conclusion:

The WEAR-AF study will explore the potential of wearable technology to transform the management of atrial fibrillation. Through this research, we aim to provide valuable data on the effectiveness of wearable ECG devices in real-world settings, offering a foundation for future innovations in digital health and personalized medicine.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Diagnosed with paroxysmal or persistent atrial fibrillation.
* Scheduled to undergo catheter ablation for atrial fibrillation.
* Able to provide informed consent.
* Willing to wear the Skiin garments (chest band or bralette) for the duration of the study (approximately 1 month pre and 6 months post-ablation).
* Have a smartphone with an Operating System compatible with the Skiin Connected Life App (Android 9+ or iOS 13+)

Exclusion Criteria:

* Adverse reaction to Skiin garments (e.g. skin allergy)

The relevant Skiin Underwear contraindications acting as exclusion criteria for this study are:

* Pacemaker and/or (ICD) implantable cardioverter defibrillator users.
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients diagnosed with atrial fibrillation (AF) who are scheduled to undergo catheter ablation. Participants must have a history of symptomatic AF and be deemed appropriate candidates for ablation by their healthcare provider. The study focuses on evaluating the use of wearable cardiac monitoring devices post-ablation, with participants being monitored for a period of 6 months to assess various outcomes related to AF recurrence, device compliance, and patient satisfaction.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Atrial Tachyarrhythmia Recurrence | 6 months post-ablation
  The primary outcome measure is the incidence of any atrial tachyarrhythmia lasting 30 seconds or longer, as detected by continuous monitoring with Skiin garments within 6 months following catheter ablation for atrial fibrillation. The occurrence of these arrhythmias will be tracked to assess the efficacy of the wearable device in detecting recurrences during the post-ablation period.

SECONDARY OUTCOMES:
Compliance with Wearable Cardiac Monitoring Device | 6 months post-ablation
  The measure of compliance will assess the proportion of time participants adhere to wearing the Skiin garments as prescribed over a 6-month period post-ablation. Compliance will be evaluated through data logs recorded by the wearable device, providing insights into participant engagement and adherence to the monitoring protocol.
Patient Satisfaction with Wearable Cardiac Monitoring Device | At the end of the 6-month monitoring period
  This outcome will evaluate patient satisfaction with the Skiin wearable cardiac monitoring device compared to traditional intermittent 14-day cardiac monitoring. Satisfaction will be measured using a validated questionnaire administered to participants at the end of the 6-month monitoring period, capturing feedback on comfort, ease of use, and overall experience with the wearable device.
Impact on Quality of Life | Baseline and 6 months post-ablation
  The impact of continuous wearable cardiac monitoring on the overall quality of life of participants post-ablation will be assessed. Quality of life will be measured using a validated tool such as the SF-36 or EQ-5D-5L at baseline and at the end of the 6-month monitoring period, with comparisons made to baseline measures and intermittent monitoring.
Time to First Recurrence of Atrial Tachyarrhythmia | From the time of ablation to the first documented recurrence within 6 months
  The time to the first documented recurrence of atrial tachyarrhythmia during continuous monitoring with Skiin garments post-ablation will be assessed. This outcome will provide insights into the efficacy of continuous monitoring in detecting arrhythmia recurrence earlier compared to traditional intermittent monitoring methods.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cheung, MD, Principal Investigator — Sunnybrook Hospital